CLINICAL TRIAL: NCT02315612
Title: Phase I Dose Escalation Study of Anti-CD22 Chimeric Receptor T Cells in Pediatric and Young Adults With Recurrent or Refractory CD22-expressing B Cell Malignancies
Brief Title: Anti-CD22 Chimeric Receptor T Cells in Pediatric and Young Adults With Recurrent or Refractory CD22-expressing B Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150029; 15-C-0029
Record Dates: First submitted 2014-12-11; First posted 2014-12-12 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-06-24

CONDITIONS: NHL; Large Cell Lymphoma; Follicular Lymphoma; ALL; B-All; B-precursor ALL; Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia; B-Non Hodgkin Lymphoma; B-NHL
Keywords: Lymphoma; Chimeric Antigen Receptor; CD-22 Expressing Tumor; ALL; Adoptive Immunotherapy; B-All; Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia; B-Non Hodgkin Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): dose escalation of CD22-CAR
  Interventions: Biological: CD22-CAR
- Arm 2 (Experimental): dose expansion of CD22-CAR
  Interventions: Biological: CD22-CAR

INTERVENTIONS:
Biological: CD22-CAR — CD22-CAR cells will be infused on Day 0 after induction chemotherapy regimen.

SUMMARY:
Background:

- One type of cancer therapy takes blood cells from a person, changes them in a lab, then gives the cells back to the person. In this study, researchers are using an anti-CD22 gene, a virus, and an immune receptor to change the cells.

Objective:

- To see if giving anti-CD22 Chimeric Antigen Receptor (CAR) cells to young people with certain cancers is safe and effective.

Eligibility:

- People ages 1-39 with a leukemia or lymphoma that has not been cured by standard therapy.

Design:

* Participants will be screened to ensure their cancer cells express the CD22 protein. They will also have medical history, physical exam, blood and urine tests, heart tests, scans, and x-rays. They may give spinal fluid or have bone marrow tests.
* Participants may have eye and neurologic exams.
* Participants will get a central venous catheter or a catheter in a large vein.
* Participants will have white blood cells removed. Blood is removed through a needle in an arm. White blood cells are removed. The rest of the blood is returned by needle in the other arm.
* The cells will be changed in a laboratory.
* Participants will get two IV chemotherapy drugs over 4 days. Some will stay in the hospital for this.
* All participants will be in the hospital to get anti-CD22 CAR cells through IV. They will stay until any bad side effects are gone.
* Participants will have many blood tests. They may repeat some screening exams.
* Participants will have monthly visits for 2-3 months, then every 3-6 months. They may repeat some screening exams.
* Participants will have follow-up for 15 years.

DETAILED DESCRIPTION:
Background:

* Adoptive cellular therapy with T cells genetically modified using viral-based vectors to express chimeric antigen receptors targeting the CD19 molecule have demonstrated dramatic clinical responses in patients with acute lymphoblastic leukemia (ALL). However, not all patients respond and CD19-negative escape has been observed following CD19 CAR therapy, as well as anti-CD19/CD3 bispecific antibody therapy. Thus, additional targets are needed.
* CD22 is a B-lineage-restricted, transmembrane phosphoglycoprotein of the Ig superfamily that is widely expressed on B-cell malignancies including 96% to 100% of pediatric Bprecursor ALL. Therefore, CD22 represents a promising target. Encouraging responses targeting CD22 with an antibody based immunoconjugate have been seen in patients, including children, with recurrent and refractory ALL. This will be the first in human testing of anti-CD22 CAR adoptive cell therapy.

Objectives:

* To determine the feasibility of producing anti-CD22 CAR cells meeting established release criteria. Complete
* To assess the safety of administering escalating doses of anti-CD22-CAR engineered T cells in children and young adults with recurrent or refractory CD22- expressing B cell malignancies following a cyclophosphamide/fludarabine preparative regimen.

Eligibility:

- Patients 3-39 years of age, at least 14.5 kg, with CD22-expressing B-cell malignancies that have recurred after or not responded to one or more standard regimens and deemed incurable by standard therapy. Patients with a history of allogeneic hematopoietic transplantation (SCT) who meet all eligibility criteria are eligible to participate. Patients previously treated with anti-CD19 CAR engineered T cells are also eligible.

Design:

* PBMC will be obtained by leukapheresis, CD3+ cells enriched and cultured in the presence of anti-CD3/-CD28 beads followed by lentiviral vector supernatant containing the anti-CD22 (M971BBz) CAR.
* On Day -4 (cell infusion is Day 0), patients will begin induction chemotherapy comprising fludarabine 25 mg/m2 on Days -4, -3, and -2 and cyclophosphamide 900 mg/m2 on day -2.
* The CD22-CAR cells will be infused on Day 0, with up to a 72h delay allowed for infusion of fresh cells or a 7 day delay if cells are cryopreserved, if needed for resolution of clinical toxicities, to generate adequate cell numbers, or to facilitate scheduling.
* A phase I cell dose escalation scheme will be performed using 3 dose levels (3 x 10(5) transduced T cells/kg; 1 x 10(6) transduced T cells/kg; and 3 x 10(6) transduced T cells/kg;). If 2/6 patients have DLT at dose level 1, safety will be evaluated in a de-escalated dose of 1 x 10(5) transduced T cells/kg (more or less 20%)). Once the maximum tolerated dose (or highest level evaluated) is reached, enrollment into an expansion cohort of a total of 83 patients at MTD will proceed to provide additional information regarding the feasibility, safety and efficacy of this treatment.
* Patients will be monitored for toxicity, response and T cell persistence as well as other biologic correlates.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patient must have a B cell ALL (inclusive of ALL blast transformation from CML) or lymphoma and must have relapsed or refractory disease after at least one standard chemotherapy regimen and one salvage regimen. In view of the PI and the primary oncologist, there must be no available alternative curative therapies and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, recurred after SCT, or have disease activity that prohibits SCT at the time of enrollment.
  2. CD22 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 80% by flow cytometry. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each patent. In general, immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood and bone marrow samples and CSF when feasible.
  3. Patients must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
  4. Greater than or equal to 3 years of age (and at least 14.5 kg) and less than or equal to 39 years of age at time of enrollment.
  5. Subjects with CNS disease are eligible, with exceptions as noted in the exclusion criteria
  6. Patients, parents/guardian(s), legally authorized representative (LAR), or durable power of attorney must be able to give consent and sign the informed consent document.
  7. Clinical performance status: Patients greater than or equal to 16 years of age: Karnofsky greater than or equal to 50%; Patients < 16 years of age: Lansky scale greater than or equal to 50%. Subjects who are unable to walk because of paralysis, but who are upright in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.
  8. Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for 12 months after receiving the preparative regimen for women and for 4 months for the same for men.
  9. Patients must have adequate organ function as described below:
* Cardiac function: Left ventricular ejection fraction greater than or equal to 45% or fractional shortening greater than or equal to 28%.
* Pulmonary function: Patients without respiratory symptoms (e.g. dyspnea at rest, known requirement for supplemental oxygen therapy) and who have an oxygen saturation greater than or equal to 92% on room air, will be eligible. For patients not meeting this criteria, pulmonary function tests will be performed to confirm that the DLCO/VA/Adj is 50% of the normal predicted value corrected for hemoglobin and alveolar volume in order to meet eligibility.(For children who are unable to cooperate for PFTs, the criterion is: No evidence of dyspnea at rest, no exercise intolerance and no requirement for supplemental oxygen therapy. )
* Hematologic function:

  * Absolute neutrophil count greater than or equal to 750/mcL
  * Platelets greater than or equal to 50,000/mcl
  * A subject will not be excluded because of pancytopenia related to disease
* Liver Function:

  * AST (SGOT)/ALT (SGPT): less than or equal to 20 x institutional upper limit of normal
  * Total bilirubin less than or equal to 2 x ULN (except in the case of subjects with documented Gilbert s disease greater than or equal to 3 x ULN)
* Renal Function: Normal creatinineCreatinine level < the maximum for age listed in the table below OR creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

  * less than or equal to 5 years old: maximum serum creatinine 0.8mg/dL
  * between 6 and 10 years old: maximum serum creatinine 1.0mg/dL
  * greater than 10 years old: maximum serum creatinine 1.2mg/dL

    10. Patients previously treated with anti-CD19 CAR or other adoptive cell therapies will be eligible if all other eligibility criteria in the expansion phase. Circulating CAR T cells must be <5% in peripheral blood.

EXCLUSION CRITERIA:

Subjects meeting any of the following criteria are not eligible for participation in the study:

1. Subjects with radiologically-detected active CNS lymphoma, leptomeningeal CNS disease or isolated CNS disease which are eligible for definitive CNS directed radiationtherapy will be excluded.
2. Hyperleukocytosis (greater than or equal to 50,000 blasts/ L) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy;
3. Pregnant or breast-feeding females
4. Recent prior therapy
5. Subjects will be excluded related to the following prior therapy criteria:

   * Systemic chemotherapy, anti-neoplastic investigational agents, or antibody based therapies <= 2 weeks (6 weeks for clofarabine or nitrosoureas) prior to apheresis with the following exception:

     --No time restriction with prior intrathecal chemotherapy, steroid therapy, hydroxyurea or ALL maintenance type chemotherapy (vincristine, 6-mercaptopurine, oral methotrexate, or a tyrosine kinase inhibitor for patients with Ph+ ALL) provided there is recovery from any acute toxic effects.
   * Radiation therapy <= 3 weeks prior to apheresis with the following exception:

     --No time restriction with radiation therapy if the volume of bone marrow treated is less than 10% and the subject has measurable/evaluable disease outside the radiation window.
   * History of allogeneic stem cell transplantation prior to apheresis that meet the following criteria:

     * Less than 100 days post-transplant
     * Evidence of active graft-versus-host disease (GVHD)
     * Taking immunosuppressive agents within 30 days prior to apheresis.
     * Less than 6 weeks post donor lymphocyte infusion (DLI)
   * History of prior CAR therapy or other adoptive cell therapies prior to apheresis that meet the following criteria:

     * Less than 30 days post-infusion
     * Circulating CAR T cells (or genetically modified cells) >=5% by flow cytometry in peripheral blood
6. HIV/HBV/HCV Infection:

   1. Seropositive for HIV antibody. (Patients with HIV are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy in the future should study results indicate effectiveness.)
   2. Positive for Hepatitis B surface antigen (HbsAG)
   3. Evidence of active HCV (evidenced by detectable HCV RNA)
7. Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject;
8. Second malignancy other than in situ carcinoma of the cervix, unless the tumor was treated with curative intent at least two years previously and subject is in remission;
9. History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study or in the manufacturing of the cells (i.e. gentamicin)

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Toxicity | End of treatment
  Number of patients who have grade 3 CRS and above
Response | 1 month, 3 months, and 6 months following CAR infusion
  Number of patients who have complete and partial remission

SECONDARY OUTCOMES:
Safety and Toxicity | 1 month, 3 months and 6 months following CAR infusion
  Number of patients who have detectable CAR cells
Objective Response (Complete + Partial Remission) | 1 month, 3 months and 6 months following CAR infusion
  The number of patients who have complete and partial remissions
CAR-T cell Persistence | 1 month, 3 months and 6 months following CAR infusion
  The number of patients who have detectable CAR cells

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Haso W, Lee DW, Shah NN, Stetler-Stevenson M, Yuan CM, Pastan IH, Dimitrov DS, Morgan RA, FitzGerald DJ, Barrett DM, Wayne AS, Mackall CL, Orentas RJ. Anti-CD22-chimeric antigen receptors targeting B-cell precursor acute lymphoblastic leukemia. Blood. 2013 Feb 14;121(7):1165-74. doi: 10.1182/blood-2012-06-438002. Epub 2012 Dec 14. PMID 23243285
- [Background] Bang S, Nagata S, Onda M, Kreitman RJ, Pastan I. HA22 (R490A) is a recombinant immunotoxin with increased antitumor activity without an increase in animal toxicity. Clin Cancer Res. 2005 Feb 15;11(4):1545-50. doi: 10.1158/1078-0432.CCR-04-1939. PMID 15746059
- [Background] Kalos M, June CH. Adoptive T cell transfer for cancer immunotherapy in the era of synthetic biology. Immunity. 2013 Jul 25;39(1):49-60. doi: 10.1016/j.immuni.2013.07.002. PMID 23890063
- [Derived] Dreyzin A, Yates B, Shalabi HN, Silbert SK, Wang HW, Yuan CM, Hoang CN, Culbert AA, Gava F, Nair MS, Giordani VM, Little L, Foley T, Nussenblatt V, Fry TJ, Stroncek DF, Highfill SL, Shah NN. 10-year experience of CD22 CAR T-cells for children and young adults with B-cell acute lymphoblastic leukemia. Blood Adv. 2025 Dec 18:bloodadvances.2025017753. doi: 10.1182/bloodadvances.2025017753. Online ahead of print. PMID 41411486
- [Derived] Silbert SK, Madan S, Holland EM, Steinberg SM, Little L, Foley T, Epstein M, Sarkisian A, Lee DW, Nikitina E, Kakumanu S, Ruppin E, Shalabi H, Yates B, Shah NN. A comprehensive analysis of adverse events in the first 30 days of phase 1 pediatric CAR T-cell trials. Blood Adv. 2023 Sep 26;7(18):5566-5578. doi: 10.1182/bloodadvances.2023009789. PMID 37486616
- [Derived] Jess J, Yates B, Dulau-Florea A, Parker K, Inglefield J, Lichtenstein D, Schischlik F, Ongkeko M, Wang Y, Shahani S, Cullinane A, Smith H, Kane E, Little L, Chen D, Fry TJ, Shalabi H, Wang HW, Satpathy A, Lozier J, Shah NN. CD22 CAR T-cell associated hematologic toxicities, endothelial activation and relationship to neurotoxicity. J Immunother Cancer. 2023 Jun;11(6):e005898. doi: 10.1136/jitc-2022-005898. PMID 37295816
- [Derived] Molina JC, Steinberg SM, Yates B, Lee DW, Little L, Mackall CL, Shalabi H, Shah NN. Factors Impacting Overall and Event-Free Survival following Post-Chimeric Antigen Receptor T Cell Consolidative Hematopoietic Stem Cell Transplantation. Transplant Cell Ther. 2022 Jan;28(1):31.e1-31.e9. doi: 10.1016/j.jtct.2021.10.011. Epub 2021 Oct 20. PMID 34687939
- [Derived] Masih KE, Ligon JA, Yates B, Shalabi H, Little L, Islam Z, Ombrello AK, Inglefield J, Nussenblatt V, Manion M, Khan J, Shah NN. Consequences of hemophagocytic lymphohistiocytosis-like cytokine release syndrome toxicities and concurrent bacteremia. Pediatr Blood Cancer. 2021 Oct;68(10):e29247. doi: 10.1002/pbc.29247. Epub 2021 Jul 26. PMID 34309174
- [Derived] Shah NN, Highfill SL, Shalabi H, Yates B, Jin J, Wolters PL, Ombrello A, Steinberg SM, Martin S, Delbrook C, Hoffman L, Little L, Ponduri A, Qin H, Qureshi H, Dulau-Florea A, Salem D, Wang HW, Yuan C, Stetler-Stevenson M, Panch S, Tran M, Mackall CL, Stroncek DF, Fry TJ. CD4/CD8 T-Cell Selection Affects Chimeric Antigen Receptor (CAR) T-Cell Potency and Toxicity: Updated Results From a Phase I Anti-CD22 CAR T-Cell Trial. J Clin Oncol. 2020 Jun 10;38(17):1938-1950. doi: 10.1200/JCO.19.03279. Epub 2020 Apr 14. PMID 32286905
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0029.html